CLINICAL TRIAL: NCT00845351
Title: Preoperative Bexarotene Treatment for Cushing's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Mary Lee Vance, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13936
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Cushing's Disease
Keywords: Cushing's
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bexarotene (Experimental): Bexarotene 300 mg/m2/day times 5 days
  Interventions: Drug: Bexarotene

INTERVENTIONS:
Drug: Bexarotene — bexarotene at 300 mg/m2/day

SUMMARY:
The objective of this pilot study is to establish the safety and tolerability of short-term therapy with bexarotene in patient's with Cushing's disease, and study the clinical, biochemical, and cellular effects of a preoperative five-day course of bexarotene in these patients before undergoing transsphenoidal surgery.

DETAILED DESCRIPTION:
Cushing's disease refers to a condition of glucocorticoid excess caused by an adrenocorticotropic hormone (ACTH) producing pituitary tumor, which account for 10-15% of all pituitary tumors. The majority of corticotroph tumors are microadenomas at the time of diagnosis, and accurate surgical and histologic identification of these tumors can be challenging. ACTH is produced in corticotroph cells within the anterior pituitary via the precursor pro-opiomelanocortin (POMC). In both physiologic and pathologic conditions the promoter for POMC is regulated by multiple transcription factors which include AP-1 and Nurr77. Retinoic acid has been shown to inhibit activation of the POMC promoter in corticotroph tumor cell culture via disruption of Nurr77 transcriptional activity. The expression of the orphan nuclear receptor termed chicken ovalbumin upstream promoter-transcription factor I (COUP-TFI) antagonizes retinoic acid signaling, and has been reported to be present in normal corticotroph cells, but lacking in adenomatous corticotroph cells in tissue culture studies. Through the retrospective analysis of 34 human corticotroph tumors we have demonstrated a consistent lack of COUP-TFI in 100% of the microadenomas that were not visible, or measured less than 5 millimeters by preoperative MRI. In total, 85% of all tumors studied showed absence of COUP-TFI. Based on in vitro data from rat and human corticotroph tumors, cells lacking COUP-TFI are vulnerable to retinoid-induced cell death via Nurr77-mediated apoptosis, an effect that is reversed by COUP-TFI gene transfection. In 2006, Castillo et al. published the results of a six-month trial which randomized 44 dogs with Cushing's disease to an RXR agonist (9-cis retinoic acid), or to ketoconazole. RXR agonist therapy outperformed ketoconazole for all endpoints, resulting in normalization of ACTH and cortisol levels in 100% of subjects that completed the study, and improved morbidity and mortality. All of the dogs treated with the RXR agonist remained in remission for the duration of the 6 to 12 month post-treatment followup.

This pilot study will involve inpatient admission to our General Clinical Research Center for 5 days prior to scheduled transsphenoidal surgery. During the five days of the study each individual will receive the RXR-agonist bexarotene at the FDA approved dose of 300 mg/m2/day. Clinical signs and symptoms of acute adrenal insufficiency will be monitored routinely throughout each 24-hour period. Baseline and twice-daily biochemical analysis for ACTH and cortisol will be performed. 24-hour urine collection for cortisol will be obtained pre-treatment and in the last 24-hours of treatment. Laboratory safety analysis will include serial comprehensive metabolic panels to monitor liver and kidney function, complete blood count to monitor for neutropenia, as well as thyroid function studies to monitor for central hypothyroidism which can develop with therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Clinical and biochemical diagnosis of Cushing's disease as established by clinical history, physical exam, and definitive biochemical testing:

  1. Persistent hypercortisolemia established by 24 hour urine free cortisol measurements
  2. Confirmation of pituitary-dependent hypercortisolemia 1. ACTH levels normal or elevated, and if clinically necessary, one of the following:

  <!-- -->

  1. Suppression of 24 hour urine free cortisol with either the 48-hour dexamethasone suppression test, or suppression of serum cortisol after an overnight high-dose (8 mg) dexamethasone suppression test -OR-
  2. Inferior Petrosal Sinus Sampling (IPSS) study
* Pituitary MRI performed within three months of enrollment
* Health status deemed appropriate for transsphenoidal surgery by the neurosurgical preoperative evaluation at the University of Virginia Pituitary Clinic

Exclusion Criteria:

* Age less than 18 or greater than 65
* Pregnant or nursing mothers
* Previous surgical, medical, or radiation therapy involving the pituitary fossa
* History of malignancy, solid or hematogenous
* History of intracranial disease, injury or intracranial surgical procedure
* Renal impairment with a GFR estimated at < 60 mL/min/1.73 m2
* History of liver disease, or baseline liver transaminase levels >50% above the upper limit of normal
* Fasting Triglycerides > 200 mg/dL
* History of pancreatitis
* Pituitary macroadenoma (> 1 cm) as measured by MRI performed within 3 months of enrollment
* Previous treatment for Cushing's disease including surgery, radiation, or medical therapy:

  1. Ketoconazole
  2. Metyrapone
  3. Aminoglutethimide
  4. Mitotane
* Oral or systemic glucocorticoid use in the last six months
* Intraarticular injection of glucocorticoids in the last year
* Current use of Ketoconazole, itraconazole, erythromycin, gemfibrozil, grapefruit juice, or other inhibitors of cytochrome P450 3A4
* Any disability or cognitive, educational, or language barriers which would inhibit the subject's ability to adequately understand the verbal and written material in the consent process despite the use of standard language translation services available through our clinic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
diurnal plasma ACTH | Days 1- 5
cortisol levels | Days 1-5
Adverse events | Days 1-5 and day two post-op

SECONDARY OUTCOMES:
clinical outcomes | Day 1-5, then at month 6 and 12, then every 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lee Vance, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States